CLINICAL TRIAL: NCT02011542
Title: Probiotics (VSL #3) for Gulf War Illness
Brief Title: Probiotic (VSL #3) for Gulf War Illness
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Original study product (VSL #3) became unavailable; change in study Collaborator and product
Sponsor: University of Utah (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ashok K. Tuteja, Professor Gastroenterology, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: W81XWH-10-1-0593
Record Dates: First submitted 2013-12-09; First posted 2013-12-13 (Estimated); Results first posted 2018-01-16 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Gulf War Illness
Keywords: Irritable Bowel Syndrome; Gulf War Illness
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo (not an active drug/ Inactive component) is given to this group
  Interventions: Drug: Placebo
- VSL #3 (Active Comparator): VSL #3 (probiotic mixture) is given to this group
  Interventions: Drug: VSL#3

INTERVENTIONS:
Drug: VSL#3 — This is a probiotic mixture
  Arms: VSL #3
Drug: Placebo — This is a pill with inactive ingredients.
  Other Names: Placebo/ Sugar pill
  Arms: Placebo

SUMMARY:
The overall objective is to determine whether VSL #3 will improve 1) intestinal symptoms of Irritable Bowel Syndrome (IBS) and 2) non-intestinal symptoms (fatigue, joint pain, insomnia, general stiffness and headache) associated with IBS. All of these symptoms are part of the Gulf War (GW) illness.

DETAILED DESCRIPTION:
Specific Aims:

Aim # 1: Determine the efficacy of VSL #3 on IBS symptoms in GW veterans.

Hypothesis: Treatment with VSL #3 compared to placebo will improve global and individual symptoms of IBS

Aim #2 Determine the efficacy VSL #3 in reducing non-intestinal symptoms of IBS (fatigue, joint pain, insomnia, general stiffness and headache).

Hypothesis: Treatment with VSL #3 compared to placebo will improve non-intestinal symptoms of IBS in GW veterans.

Aim #3 Determine whether changes in gut flora and plasma cytokines correlate with treatment response in GW veterans.

ELIGIBILITY:
Inclusion Criteria:

1. First GW veterans, Men and women age 35-75 years,
2. Rome III criteria for IBS and two or more of the non-intestinal symptoms (chronic-once a week or more often-fatigue, joint pains, insomnia, general stiffness, and headache)
3. Symptoms of > 6 months duration,
4. No significant findings on physical examination, Complete Blood Count (CBC) and clinical chemistry panel.
5. Normal gross appearance of the colonic mucosa other than erythema and polyps
6. Negative Tissue transglutaminase (TTG) for celiac disease,
7. Normal thyroid function.
8. Veterans with psychological disorders will not be excluded but will be identified for sub-group analysis.
9. Stable medication regimen for more than a month

Exclusion Criteria:

1. Current evidence of any lower gastrointestinal disorder such as celiac disease or inflammatory bowel disease
2. History of/or presence of systemic malignancy (patients with skin and other cancers in remission for more than 5 years are allowed in the study
3. Clinically significant chronic disease: HIV, cardiac, pulmonary, hepatic or renal dysfunction.
4. Presence of Giardia antigen, and Clostridium difficile toxin in stool,
5. Abnormal blood test for thyroid stimulating hormone, tissue transglutaminase antibody
6. Current effects of drug or alcohol abuse
7. Investigator perception of patient's inability to comply with study protocol
8. Recent change in gastrointestinal medications
9. Use of any antibiotic in the last 1 months
10. Positive pregnancy test
11. Subject is currently participating in another research protocol that could interfere or influence the outcome measures of the present study.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- George E Wahlen VA Medical Center, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study is ongoing; information on enrolled participant arm assignment is blinded, therefore these arms/groups are combined
Groups:
- VSL #3 or Placebo: Study participants enrolled into the VSL #3 arm or the Placebo arm
Period: Overall Study
Arm/Group | VSL #3 or Placebo
Started | 30
Completed | 29
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Clinical trial is ongoing; change in collaborator and investigational product required new study registration. Clinical trial results for all participants will be reported upon study completion in record NCT03078530.
Arm/Group | VSL #3 or Placebo
Number analyzed (Participants) | 0
Age, Continuous
Sex: Female, Male

OUTCOME MEASURES:

1. Primary Outcome: Improvement in the Bowel Symptom Scale (BSS) From Baseline
Description: Efficacy of VSL #3 in Irritable Bowel Syndrome (IBS) related symptoms in Gulf War illness is measured using BSS at 2, 4, 6, 8 wks
Time Frame: 8 weeks
Population: as for baseline characteristics
Arm/Group | VSL #3 or Placebo
Number analyzed (Participants) | 0

2. Secondary Outcome: Change in Chronic Fatigue (1-5 Scale) From Baseline
Description: Efficacy of VSL #3 in reducing non-intestinal symptoms of IBS is measured using chronic fatigue scale at 2,4,6,8, weeks
Time Frame: 8 weeks
Population: as for baseline characteristics
Arm/Group | VSL #3 or Placebo
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Clinical trial is ongoing; change in collaborator and investigational product required new study registration. Clinical trial results for all participants will be reported upon study completion in record NCT03078530.
Arm/Group | VSL #3 or Placebo
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Clinical trial is ongoing; change in collaborator and investigational product required new study registration. Clinical trial results for all participants will be reported upon study completion in record NCT03078530.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No